CLINICAL TRIAL: NCT01872143
Title: Non-invasive Brain Stimulation for the Treatment of Psychiatric Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, giordano d'urso, MD, PhD, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61/10 (Ethical Committee)
Record Dates: First submitted 2013-05-16; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transcranial Direct Current Stimulation (Experimental): daily or twice-a-day administration of transcranial Direct Current Stimulation
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — daily or twice-a-day administration of transcranial Direct Current Stimulation from a minimum of 10 session to a maximum of 20

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS) is effective in the treatment of psychiatric disorders in which available treatments are either ineffective or not tolerated

DETAILED DESCRIPTION:
Depending on the specific psychiatric disorder, inhibitory or stimulating neuromodulation will be applied over the cortical region of interest, found according to the relevant scientific publication on neurophysiology of psychiatric disorders

ELIGIBILITY:
Inclusion Criteria:

* a psychiatric disorder in which available treatment are either ineffective or not tolerated

Exclusion Criteria:

* implantable active devices

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Psychiatric rating scales scores at immediate post-treatment and at one-month and at three-month follow-up visits | Time points: T0=baseline; T1=immediate post-treatment; T2=one-month follow-up visit; T3=3-months follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: giordano d'urso, MD, PhD, Principal Investigator — AOU "Federico II" of Naples
Locations (1):
- AOU "Federico II" of Naples, Naples, Italy